CLINICAL TRIAL: NCT03331874
Title: Reflectance Confocal Microscopy to Diagnose Basal Cell Carcinoma
Brief Title: RCM to Diagnose BCC - Reflectance Confocal Microscopy to Diagnose Basal Cell Carcinoma
Acronym: RCM-1
Status: Completed | Type: Observational
Sponsor: Julie Dawson (Other)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 206698(59-03-16)
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Basal Cell Carcinoma
Keywords: confocal; basal; carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Basal Cell Carcinoma: Diagnosis of Basal Cell Carcinoma by Reflectance confocal microscopy
  Interventions: Diagnostic Test: Reflectance Confocal Microscopy

INTERVENTIONS:
Diagnostic Test: Reflectance Confocal Microscopy — In-vivo microscope

SUMMARY:
Basal cell carcinoma (BCC) is the commonest non melanoma skin cancer in the UK and its incidence is rising. The Norfolk and Norwich University Hospital Foundation Trust (NNUHFT) see and excise approximately 3,000 new cases of BCC each year. Many of these patients have a biopsy to confirm their diagnosis before being listed for surgical excision. In vivo reflectance confocal microscopy (RCM) involves using a machine which can examine the upper layers of the skin non invasively.

In clinically suspicious lesions, the Investigators will use RCM prior to biopsy with the aim of demonstrating that RCM can accurately diagnose BCC. The aim of this study is to determine the feasibility and utility of using RCM for the diagnosis of BCC in the NHS setting, thereby shortening the patient pathway and effectively using limited public resources. If the Investigators' study shows that RCM can accurately diagnose BCC in these patients then this would prevent the need for biopsy as a routine in these patients.

DETAILED DESCRIPTION:
Patients will be recruited from the outpatient clinics of the Departments of Dermatology and Plastic Surgery at the Norfolk and Norwich University Hospital Foundation Trust. These will be patients who have been assessed in clinic by a consultant dermatologist or consultant plastic surgeon. They will be suspected of having a BCC on the head and neck region. Clinical and dermoscopic (a dermatoscope is a hand held microscope) images will be taken by the Medical Illustration at NNUHFT as part of their routine standard of care. Patients will be invited to participate in the trial and provided with a patient information leaflet. They will be given sufficient time to review the information sheet and ask questions. Patients will be consented to having reflectance confocal microscopy performed of the target lesion before undergoing biopsy for histology. These patients would be having photographs, including dermoscopic images, and a biopsy as part of their standard of care prior to their final treatment being determined - the only additional intervention is examination with the confocal microscope.

The images taken of the tumour by the reflectance confocal microscope will be anonymised. These images will then be examined by a different in house dermatologist who has undergone training in examining confocal images. The images will also be sent to a dermatologist in Modena, Italy who is experienced in interpreting confocal microscopic images - both of these dermatologists will be blinded as to the patient's history and the results of the punch biopsy.

The biopsies will undergo routine processing in our histopathology laboratory as normal and will be analysed by a pathologist who will be unaware of the findings on confocal microscopy.

The patients will undergo one additional intervention over-and-above their standard investigation and treatment pathway. The treatment pathway for the patients will not be lengthened or shortened by their participation.

ELIGIBILITY:
Inclusion Criteria: Patients 18 years or older with a suspected diagnosis of BCC of the head and neck region.

-

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See Above
Sampling Method: Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Specificity & Sensitivity of RCM in diagnosing BCC compared to standard histology | 18 months
  Specificity & Sensitivity of RCM in diagnosing BCC compared to standard histology

SECONDARY OUTCOMES:
Inter- & intra-observer agreement in assessing RCM images | 18 months
  Inter- & intra-observer agreement in assessing RCM images

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Garioch, Dr, Principal Investigator — Consultant Oncologist
Locations (1):
- Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levell NJ, Igali L, Wright KA, Greenberg DC. Basal cell carcinoma epidemiology in the UK: the elephant in the room. Clin Exp Dermatol. 2013 Jun;38(4):367-9. doi: 10.1111/ced.12016. Epub 2013 Mar 18. PMID 23496262
- [Background] Sauermann K, Gambichler T, Wilmert M, Rotterdam S, Stucker M, Altmeyer P, Hoffmann K. Investigation of basal cell carcinoma [correction of carcionoma] by confocal laser scanning microscopy in vivo. Skin Res Technol. 2002 Aug;8(3):141-7. doi: 10.1034/j.1600-0846.2002.20345.x. PMID 12236882
- [Background] Gonzalez S, Tannous Z. Real-time, in vivo confocal reflectance microscopy of basal cell carcinoma. J Am Acad Dermatol. 2002 Dec;47(6):869-74. doi: 10.1067/mjd.2002.124690. PMID 12451371
- [Background] Goldgeier M, Fox CA, Zavislan JM, Harris D, Gonzalez S. Noninvasive imaging, treatment, and microscopic confirmation of clearance of basal cell carcinoma. Dermatol Surg. 2003 Mar;29(3):205-10. doi: 10.1046/j.1524-4725.2003.29050.x. PMID 12614409
- [Background] Marra DE, Torres A, Schanbacher CF, Gonzalez S. Detection of residual basal cell carcinoma by in vivo confocal microscopy. Dermatol Surg. 2005 May;31(5):538-41. doi: 10.1111/j.1524-4725.2005.31157. PMID 15962737
- [Background] Nori S, Rius-Diaz F, Cuevas J, Goldgeier M, Jaen P, Torres A, Gonzalez S. Sensitivity and specificity of reflectance-mode confocal microscopy for in vivo diagnosis of basal cell carcinoma: a multicenter study. J Am Acad Dermatol. 2004 Dec;51(6):923-30. doi: 10.1016/j.jaad.2004.06.028. PMID 15583584
- [Background] Longo C, Farnetani F, Ciardo S, Cesinaro AM, Moscarella E, Ponti G, Zalaudek I, Argenziano G, Pellacani G. Is confocal microscopy a valuable tool in diagnosing nodular lesions? A study of 140 cases. Br J Dermatol. 2013 Jul;169(1):58-67. doi: 10.1111/bjd.12259. PMID 23374159
- [Background] Gerger A, Koller S, Weger W, Richtig E, Kerl H, Samonigg H, Krippl P, Smolle J. Sensitivity and specificity of confocal laser-scanning microscopy for in vivo diagnosis of malignant skin tumors. Cancer. 2006 Jul 1;107(1):193-200. doi: 10.1002/cncr.21910. PMID 16615102
- [Background] Eichert S, Mohrle M, Breuninger H, Rocken M, Garbe C, Bauer J. Diagnosis of cutaneous tumors with in vivo confocal laser scanning microscopy. J Dtsch Dermatol Ges. 2010 Jun;8(6):400-10. doi: 10.1111/j.1610-0387.2010.07333.x. Epub 2010 Feb 5. English, German. PMID 20141551
- [Background] Guitera P, Menzies SW, Longo C, Cesinaro AM, Scolyer RA, Pellacani G. In vivo confocal microscopy for diagnosis of melanoma and basal cell carcinoma using a two-step method: analysis of 710 consecutive clinically equivocal cases. J Invest Dermatol. 2012 Oct;132(10):2386-2394. doi: 10.1038/jid.2012.172. Epub 2012 Jun 21. PMID 22718115
- [Background] Peppelman M, Wolberink EA, Blokx WA, van de Kerkhof PC, van Erp PE, Gerritsen MJ. In vivo diagnosis of basal cell carcinoma subtype by reflectance confocal microscopy. Dermatology. 2013;227(3):255-62. doi: 10.1159/000354762. Epub 2013 Oct 18. PMID 24158236
- [Background] Castro RP, Stephens A, Fraga-Braghiroli NA, Oliviero MC, Rezze GG, Rabinovitz H, Scope A. Accuracy of in vivo confocal microscopy for diagnosis of basal cell carcinoma: a comparative study between handheld and wide-probe confocal imaging. J Eur Acad Dermatol Venereol. 2015 Jun;29(6):1164-9. doi: 10.1111/jdv.12780. Epub 2014 Oct 22. PMID 25338750